CLINICAL TRIAL: NCT06511830
Title: The Effectiveness of Detecting Plaque on Tooth Surfaces Using Traditional and Artificial Intelligence Monitoring
Brief Title: Effectiveness of Plaque Score Detection Techniques
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0341-24-FB
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dental Monitoring images — Dental Monitoring is a series of intraoral photos that will be taken and assessed to determine the subject's dental plaque levels.

SUMMARY:
This study investigates the similarity between microbial plaque scores when assessing the entire dentition versus select teeth. The hypothesis posits that plaque buildup on single teeth mirrors that of the entire mouth, facilitating efficient plaque data collection and generalized deductions. Additionally, the research explores the potential of Dental Monitoring© photos in accurately identifying plaque indexes, aiming to enhance plaque evaluation efficiency in dental appointments. The null hypothesis suggests no significant difference between full dentition plaque scores and selected teeth. Results may streamline plaque tracking in patient appointments and enable remote monitoring, potentially detecting plaque accumulation issues earlier.

DETAILED DESCRIPTION:
Following the obtainment of participant consent, data will be collected during participant's routine prophylaxis appointment or during designated clinic time open for participants to volunteer. Utilizing a scan box provided by Dental Monitoring©, a scan (series of intra-oral images) will be taken of the participant's dentition. The scan will be taken once before disclosing solution (erythrosine) is introduced to the dentition and once after.

The disclosing solution will allow for visualization of plaque. The presence of plaque on all teeth surfaces will be recorded using the O'Leary Plaque Index. No procedures (other than the intra-oral photos), interventions, evaluations or tests will be performed more frequently than they would be if the participant was not participating in the research. The only participant demographic information that will be recorded for this study is age.

Participants who opt to come in voluntarily for only data collection will not receive a prophylaxis. Their plaque information will be collected, and they will be dismissed.

Oversight procedures in place: The Scan Boxes will be utilized by the investigators to take intra-oral photographs of each patient's dentition. These will be sterilized between each participant and stored in the College of Dentistry's clinic lockers when not in use.

ELIGIBILITY:
Inclusion Criteria:

* 19-85 years old
* Patient at the University of Nebraska Medical Center (UNMC) College of Dentistry
* One molar, premolar or canine pe quadrant

Exclusion Criteria:

* No permanent dental devices (braces, splints)
* Less than 20 non-restored teeth present in the dentition

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be routine patients at the UNMC College of Dentistry clinics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence of Visibly Detectable Plaque | Baseline
  The presence of dental plaque will be determined by visual presence or absence of dental plaque at 6 sites per tooth. The presence of dental plaque is reported as a percentage of tooth surfaces with visibly detectable plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Killeen, DDS, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center Dental College, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No